CLINICAL TRIAL: NCT02380703
Title: Aggression Prevention Training for Caregivers of Persons With Dementia (APT)
Acronym: APT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mark Kunik, M.D., M.P.H., Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-33720; R01NR014657-01A1 (NIH)
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Dementia; Pain; Alzheimer's Disease; Aggression; Depression; Interpersonal Relations
Keywords: aggression; dementia; Alzheimer's disease; pain; depression; caregiver; behavioral health; counseling
MeSH Terms: conditions — Dementia; Pain; Alzheimer Disease; Aggression; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aggression Prevention Training (APT) (Experimental): APT will use active learning tools, including didactics, role-playing, and multimedia (eg, books and DVDs) to educate and provide skill training for the caregiver. The 6-8 modules in the intervention will include 4 core modules that address 4 main aggression risk factors: a) recognizing pain, b) treating pain, c) increasing pleasant activities, and d) improving patient-caregiver communication. Caregivers can select 2 to 3 additional elective sessions; elective selection is guided by the needs of the dyad to further enhance skills related to these core topics. Sessions will take place in the patient's home.
  Interventions: Behavioral: Aggression Prevention Training (APT)
- Enhanced Usual Primary Care (EU-PC) (Placebo Comparator): EU-PC provides the patient and caregiver educational materials on pain, notifies the primary care provider of the PWD's level of pain and depression, and provides 8 weekly supportive telephone calls to caregivers.
  Interventions: Other: Enhanced Usual Primary Care (EU-PC)

INTERVENTIONS:
Behavioral: Aggression Prevention Training (APT)
  Arms: Aggression Prevention Training (APT)
Other: Enhanced Usual Primary Care (EU-PC)
  Arms: Enhanced Usual Primary Care (EU-PC)

SUMMARY:
This study will evaluate whether a home-based targeted education and skill training (Aggression Prevention Training or APT) will reduce aggression in persons with dementia (PWD) and pain/pain-related features more than usual care plus supportive telephone calls. Half of the participants will receive APT and half will receive supportive telephone calls.

DETAILED DESCRIPTION:
Eighty percent of PWD have behavioral or psychological disturbances, including 40% that are aggressive behaviors. The prevalence of pain in PWD is about 60%, and it is a strong predictor of aggression. The biopsychosocial model of pain posits that pain is bidirectionally related to psychological factors (ie, depression) and social support factors (ie, quality of caregiver/PWD relationship) in addition to biological factors. Thus, depression and quality of the caregiver/PWD relationship can be seen as pain-related features. Caregivers are ideally suited to help address pain, depression, and the caregiver/PWD relationship, thus preventing the development of aggression; but they need tools to assist them in identifying and managing these symptoms.

Prior studies of aggression treatment have not examined using a preventive strategy to decrease incidence of aggression in persons with dementia (PWD). Almost all studies have examined use of pharmacologic interventions following development of aggression.This 5-year randomized controlled trial based on the Unmet Needs Model will focus on preventing aggression in PWD with pain and pain-related features by providing the caregiver with targeted education and skill training. PWD and their caregivers will be randomized to APT or to an enhanced usual primary care condition (EU-PC). APT will use active learning tools, including didactics, role-playing, and multimedia [eg, books and digital versatile discs (DVDs)] to educate and provide skill training for the caregiver. The 6-8 modules in the intervention will include 4 core modules that address 4 main aggression risk factors: a) recognizing pain, b) treating pain, c) increasing pleasant activities, and d) improving patient-caregiver communication. Caregivers can select 2 to 3 additional elective sessions; elective selection is guided by the needs of the dyad to further enhance skills related to these core topics. EU-PC provides the patient and caregiver educational materials on pain, notifies the primary care provider of the PWD's level of pain and depression, and provides 8 weekly supportive telephone calls to caregivers. PWD and caregiver outcomes will be collected at baseline, 3, 6 and 12 months.

Data analysis will include both univariate descriptive statistics and inferential statistics, including regression models, repeated measure modeling and Cox proportional hazards models.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of dementia
2. Clinically significant pain, depression, or caregiver/patient relationship difficulties (either self-report or caregiver proxy-report).
3. Receives care from Baylor College of Medicine Geriatric Medicine Associates or Alzheimer's Disease and Memory Disorders Center, or Kelsey Seybold Clinics
4. Has an informal caregiver willing to participate in the study who sees the patient at least 8 hours/week and at least twice/week
5. Speaks English
6. Lives within a 40-mile radius of the coordinating center

Exclusion Criteria:

1. Advanced dementia based on inability to complete the Mental Impairment Screen-Telephone Version or a Functional Assessment Staging Tool score > 6.
2. History of aggression during the one month prior to screening or baseline
3. Resides in a long-term care facility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Kunik, M.D., Ph.D., Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No
The information generated in this proposal aims to prevent the development of aggression in persons with dementia. Clinician and participant manuals are developed for the intervention and will be widely shared through abstracts, presentation, publication and personal communication if the intervention is efficacious. In addition, if the intervention is found to be evidence-based, we will pursue placement on the websites of:
  1) Substance Abuse and Mental Health Services Administration (SAMHSA) National Registry for Evidence-based Programs and 2) Rosalynn Carter Institute for Caregiving (RCI) Caregiver Intervention Database. Information about the study will also be available to interested investigators through NIH CRISP, and the Baylor College of Medicine Section of Health Services Research website. Requests to use the information will be considered on a case-by-case basis, following written request to the principal investigator.

REFERENCES:
- [Derived] Sibley AA, Shrestha S, Lipovac-Dew M, Kunik ME. Examining Depression Symptoms With/Without Coexisting Anxiety Symptoms in Community-Dwelling Persons With Dementia. Am J Alzheimers Dis Other Demen. 2021 Jan-Dec;36:1533317521990267. doi: 10.1177/1533317521990267. PMID 33530695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2,230 persons with dementia (PWD) were contacted for telephone screening; 253 were interested and eligible for the study
Pre-assignment Details: 239 signed written informed consent and 233 completed baseline assessments (5 were lost and 1 withdrew after signing consent); 4 were excluded at baseline due to the presence of aggression in the 3 months prior to baseline based on Cohen-Mansfield Agitation Inventory (CMAI); 1 participant withdrew prior to randomization; 228 participants were randomly assigned to a study arm (114 in each group).
Groups:
- Aggression Prevention Training (APT): APT will use active learning tools, including didactics, role-playing, and multimedia [eg, books and digital video disc (DVDs)] to educate and provide skill training for the caregiver. The 6-8 modules in the intervention will include 4 core modules that address 4 main aggression risk factors: a) recognizing pain, b) treating pain, c) increasing pleasant activities, and d) improving patient-caregiver communication. Caregivers can select 2 to 3 additional elective sessions; elective selection is guided by the needs of the dyad to further enhance skills related to these core topics. Sessions will take place in the patient's home.
  Aggression Prevention Training (APT)
- Enhanced Usual Primary Care (EU-PC): EU-PC provides the patient and caregiver educational materials on pain, notifies the primary care provider of the PWD's level of pain and depression, and provides 8 weekly supportive telephone calls to caregivers.
  Enhanced Usual Primary Care (EU-PC)
Period: Overall Study
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Started (This is the number of PWD assigned to each arm.) | 114 | 114
Month 3 (This is the number of PWD who reached the Month 3 assessment window.) | 104 | 109
Month 6 (This is the number of PWD who reached the Month 6 assessment window.) | 102 | 107
Month 12 (This is the number of PWD who reached the Month 12 assessment window.) | 99 | 100
Completed (This is the number of PWD who completed the Month 12 assessment.) | 78 | 78
Not Completed | 36 | 36
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Lost to Follow-up | 12 | 12
Not completed — Caregiver death | 1 | 0
Not completed — Person with dementia (PWD) death | 7 | 8
Not completed — Entered Long-term Care | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Aggression Prevention Training (APT): APT will use active learning tools, including didactics, role-playing, and multimedia (eg, books and DVDs) to educate and provide skill training for the caregiver. The 6-8 modules in the intervention will include 4 core modules that address 4 main aggression risk factors: a) recognizing pain, b) treating pain, c) increasing pleasant activities, and d) improving patient-caregiver communication. Caregivers can select 2 to 3 additional elective sessions; elective selection is guided by the needs of the dyad to further enhance skills related to these core topics. Sessions will take place in the patient's home.
  Aggression Prevention Training (APT)
- Total: Total of all reporting groups
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC) | Total
Number analyzed (Participants) | 114 | 114 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.98 (9.16) | 78.31 (8.75) | 78.15 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 66 | 65 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 78 | 75 | 153
  Black | 24 | 24 | 48
  Hispanic | 9 | 12 | 21
Individual with Dementia-reported Overall Pain [Mean (Standard Deviation); unit: units on a scale] — The Philadelphia Geriatric Pain Intensity Scale will be administered to the PWD to measure pain. It consists of 4 items assessing the extent to which the PWD has been bothered by pain over the past several weeks--at present, when pain was at its worst, when pain was at its least, and overall. These items are rated on a 0- to 5-point Likert scale (not at all to extremely). A fifth item asks for number of days per week that pain was really bad, and a sixth asks for a rating of how much pain has interfered with day-to-day activities. We report only on the item about overall pain.
  units on a scale | 1.38 (1.12) | 1.13 (1.24) | 1.25 (1.18)
Caregiver-reported Overall Pain [Mean (Standard Deviation); unit: units on a scale] — The Philadelphia Geriatric Pain Intensity Scale will be administered to the caregiver to measure their report of PWD pain. It consists of 4 items assessing extent to which the caregiver feels the PWD has been bothered by pain over the past several weeks--at present, when pain was at its worst, when pain was at its least, and overall. Items are rated on a 0- to 5-point Likert scale (not at all to extremely). A 5th item asks for number of days per week pain was really bad, and a 6th asks for a rating of how much pain interfered with day-to-day activities. We report only on the overall pain item.
  units on a scale | 1.44 (1.11) | 1.16 (1.12) | 1.30 (1.12)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — The 30-item GDS will be administered to the caregiver to measure depression. Items are answered with Yes/No. Total score ranges from 0-30. A score of 11 or greater is a possible indicator of depression.
  units on a scale | 11.88 (6.25) | 11.10 (6.48) | 11.49 (6.36)
Mutuality Scale [Mean (Standard Deviation); unit: units on a scale] — The Mutuality Scale and is a 15-item instrument measuring the positive quality of the relationship between caregiver and care receiver. Questions are answered by the caregiver on a 5-point Likert-type scale (0=never, 4=a great deal). Its 4 subscales represent domains of shared values, affective closeness, shared pleasurable activities and reciprocity. The total score ranges from 0-4 and is the sum of individual items divided by the number of items answered. High scores indicate a relationship characterized by communication, shared pleasurable activities, common values, and reciprocity.
  units on a scale | 2.93 (0.79) | 3.05 (0.76) | 2.99 (0.78)
Zarit Burden Inventory [Mean (Standard Deviation); unit: units on a scale] — The Zarit Burden Interview is a 22-item instrument measuring perceived impact of caregiving on the caregiver's financial status, physical status, physical health, emotional health, and social activities. Questions are answered on a 5-point Likert-type scale (0=never, 4=nearly always). The total scale score ranges from 0-88.
  units on a scale | 27.77 (15.03) | 27.00 (13.29) | 27.39 (15.13)
Positive Aspects of Caregiving [Mean (Standard Deviation); unit: units on a scale] — The 9-item Positive Aspects of Caregiving Scale presents statements about a caregiver's mental or affective state in the context of the caregiving experience. Responses are provided on a 5-point agree/disagree scale and designed to assess perception of benefits within the caregiving context, such as feeling useful, feeling appreciated, and finding meaning. Higher scores (range 9-45) represent more positive appraisals.
  units on a scale | 24.18 (9.00) | 23.88 (9.54) | 24.03 (9.25)
Revised Memory and Behavior Checklist (RMBC) - Total Frequency [Mean (Standard Deviation); unit: units on a scale] — Revised Memory and Behavior Checklist (RMBCL) is a 24-item informant-based measure of observable behavior problems in PWD, including memory-related, disruptive, and depressive behaviors. Scores are computed for the presence/absence of each problem first and then for caregiver "reaction" or the extent to which caregivers were bothered or distressed by each behavior (0-4). Total score is the sum of reaction scores for all endorsed behaviors. Possible range is 0-96. A higher score indicates a worse outcome.
  units on a scale | 8.13 (3.79) | 7.56 (3.43) | 7.85 (3.62)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aggression as Per the Cohen Mansfield Agitation Inventory, Aggression Subscale
Description: Aggression is measured on a 7-point Likert scale for frequency and a 5-point Likert scale for disruptiveness. Aggression is considered present if a participant scores over one on both frequency (more than never) and disruptiveness (at least a little) on any of 13 aggressive behaviors, including spitting, verbal aggression, hitting, kicking, grabbing, pushing, throwing, biting, scratching, hurting self/others, destroying property, or making inappropriate verbal or physical sexual advances.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
Participants | 29 | 23
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); Sample-size calculations were performed, based on the ability to detect a small-to-moderate difference (Cohen's h = 0.4) in rate of aggression onset over a 1-year period between APT and EU-PC, assuming 80% power and a type I error rate of 5%. Given an anticipated rate of aggression onset over 1 year of 37% for EU-PC, an ES of h = 0.4 allows detection of aggression onset in APT as high as 19%. Given this effect size and up to 10% attrition, our goal was to include 220 total participants; Test type: Superiority; p = 0.29, Regression, Cox — For participants who dropped out, their time until study attrition was used as the exposure period; and they were carried forward as part of the overall incidence count; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.78 to 2.32]
Statistical Analysis 2: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); Test type: Equivalence — Examination of whether the presence of aggression is equivalent between APT and EU-PC; p = 0.27, Chi-squared — Association between presence of aggression and condition (APT vs EU-PC); X2(1) = 1.21; Difference in frequencies = 1.21

2. Secondary Outcome: Caregiver Burden--Zarit Burden Interview
Description: The Zarit Burden Interview is a 22-item instrument measuring perceived impact of caregiving on the caregiver's financial status, physical status, physical health, emotional health, and social activities. Questions are answered on a 5-point Likert-type scale (0=never, 4=nearly always). The total scale score ranges from 0-88.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 26.12 (14.72) | 28.37 (16.27)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); Differences between APT and EU-PC in change over time (baseline, and 3, 6 and 12 months) for our secondary outcomes were evaluated using individual linear growth curve models (SAS Proc Mixed, SAS Institute, Inc., Cary, NC) with an autoregressive covariance structure type. The main interest was the interaction between group (APT vs EU-PC) and time; Test type: Superiority; p = 0.19, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 1.59 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

3. Secondary Outcome: Positive Caregiving Attributes--Positive Aspects of Caregiving Scale
Description: The 9-item Positive Aspects of Caregiving Scale presents statements about a caregiver's mental or affective state in the context of the caregiving experience. Responses are provided on a 5-point agree/disagree scale and designed to assess perception of benefits within the caregiving context, such as feeling useful, feeling appreciated, and finding meaning. Higher scores (range 9-45) represent more positive appraisals.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 25.87 (8.46) | 25.00 (9.53)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.06, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 2.43 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

4. Secondary Outcome: Behavior Problems--Revised Memory and Behavior Checklist
Description: Revised Memory and Behavior Checklist (RMBCL) is a 24-item informant-based measure of observable behavior problems in PWD, including memory-related, disruptive, and depressive behaviors. Scores are computed for the presence/absence of each problem first and then for caregiver "reaction" or the extent to which caregivers were bothered or distressed by each behavior (0-4). Total score is the sum of reaction scores for all endorsed behaviors. Possible range is 0-96. A higher score indicates a worse outcome.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 7.86 (4.37) | 7.51 (4.08)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.80, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 0.33 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

5. Secondary Outcome: Pain--Philadelphia Geriatric Pain Intensity Scale (Overall Pain as Reported by the PWD)
Description: The Philadelphia Geriatric Pain Intensity Scale will be administered to the PWD to measure pain. It consists of 4 items assessing the extent to which the PWD has been bothered by pain over the past several weeks--at present, when pain was at its worst, when pain was at its least, and overall. These items are rated on a 0- to 5-point Likert scale (not at all to extremely). A fifth item asks for number of days per week that pain was really bad, and a sixth asks for a rating of how much pain has interfered with day-to-day activities. We report only on the item about overall pain.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 1.19 (1.14) | 1.12 (1.19)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.89, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 0.21 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

6. Secondary Outcome: Depression--Geriatric Depression Screen (GDS), Caregiver Version
Description: The 30-item GDS will be administered to the caregiver to measure depression. Items are answered with Yes/No. Total score ranges from 0-30. A score of 11 or greater is a possible indicator of depression.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 12.06 (6.98) | 11.43 (7.42)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.22, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 1.48 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

7. Secondary Outcome: Caregiver-Patient Relationship Quality--Mutuality Scale
Description: The Mutuality Scale and is a 15-item instrument measuring the positive quality of the relationship between caregiver and care receiver. Questions are answered by the caregiver on a 5-point Likert-type scale (0=never, 4=a great deal). Its 4 subscales represent domains of shared values, affective closeness, shared pleasurable activities and reciprocity. The total score ranges from 0-4 and is the sum of individual items divided by the number of items answered. High scores indicate a relationship characterized by communication, shared pleasurable activities, common values, and reciprocity.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 2.91 (0.85) | 2.99 (0.78)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.77, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 0.38 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

8. Secondary Outcome: Pain--Philadelphia Geriatric Pain Intensity Scale (Overall Pain as Reported by the Caregiver)
Description: The Philadelphia Geriatric Pain Intensity Scale will be administered to the caregiver to measure caregiver report of PWD pain. It consists of 4 items assessing the extent to which the the caregiver feels the PWD has been bothered by pain over the past several weeks--at present, when pain was at its worst, when pain was at its least, and overall. These items are rated on a 0- to 5-point Likert scale (not at all to extremely). A fifth item asks for number of days per week that pain was really bad, and a sixth asks for a rating of how much pain has interfered with day-to-day activities. We report only on the item about overall pain.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
Number analyzed (Participants) | 114 | 114
units on a scale | 1.48 (1.07) | 1.20 (1.10)
Statistical Analysis 1: Comparison: Aggression Prevention Training (APT) vs Enhanced Usual Primary Care (EU-PC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.64, Mixed Models Analysis — P value for interaction between treatment arm and time; F-statistic = 0.56 — Interaction between time and treatment arm: Numerator df = 3, denominator df = 510

ADVERSE EVENTS:
Time Frame: Serious Adverse Events data were collected through the end of the study (Month 12). All events were considered unrelated to the study.
Description: This is a minimal risk behavioral intervention. Non-serious adverse events were not collected.
Arm/Group | Aggression Prevention Training (APT) | Enhanced Usual Primary Care (EU-PC)
All-Cause Mortality (participants affected / at risk) | 7/114 | 7/114
Serious Adverse Events (participants affected / at risk) | 15/114 | 18/114
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggression Prevention Training (APT) (N=114) | Enhanced Usual Primary Care (EU-PC) (N=114)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 3 (3)
Hospitalization (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hospitalization (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 0 (0) | 3 (3)
Hospitalization (Renal and urinary disorders) | 2 (2) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 5 (5) — No information on cause of death
Death (Cardiac disorders) | 1 (1) | 0 (0)
Death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (Nervous system disorders) | 1 (1) | 1 (1)
Death (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02380703/Prot_SAP_000.pdf